CLINICAL TRIAL: NCT04354792
Title: Asymptomatic SARS- CoV2 Infection Among Healthcare Workers in Three University Hospitals: A Cross Sectional Study.
Brief Title: Asymptomatic COVID-19 Infection Among Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mukhtar, professor of anesthesia and intensive care, Kasr El Aini Hospital
Other Study IDs: N-31-2020
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Immunologic Activity Alteration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum SARsCOV-2 IGg to assess immunological state of HCWs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum SARs COV 2 IGg screening in health care workers — Blood samples will be collected from the enrolled HCWs. Sample collection, processing, and laboratory testing will follow guidance from the World Health Organization

SUMMARY:
To assess the seroprevalence of SARS-CoV-2 IgG in Health care workers in three University Hospitals

DETAILED DESCRIPTION:
The proposed study is a cross sectional study that will be carried out among HCWs in three University hospitals namely Kasr Alaini , Ain Shams , and Zagazeg Hospitals, employing a quantitative survey.

II-Study population Participants will be the HCWs at great risk of getting an infection which include those who are in direct contact with respiratory secretions.

Inclusion criteria Age: From 25 to 60 years old Department: physicians and nurses from the operating room, critical care department, emergency department, pulmonology department.

The potential participants will be given an information sheet and time to review this information before informed consent is sought. After the potential participants have agreed to be enrolled in the study, an informed consent will be obtained by the Investigator.

III- Procedures and Data collection:

Serum Collection and Interview A- Detecting Serum IgG against SARS-CoV2

Blood samples will be collected from the enrolled HCWs. Sample collection, processing, and laboratory testing will follow guidance from the World Health Organization.(5) The sensitivity and specificity reported by the manufacturer for IgM are 88.2% and 99.0% respectively, and for IgG are 97.8% and 97.9%.

B- Structured Interview questionnaire

A structured - interview questionnaire using closed ended question format will be used to obtain information on:

1. Socio-demographic characteristics of the interviewees asking about age, sex, residence, education, occupation, department, Job title, hospital name, medical experience in years, marital status, living with family, and having children or not.
2. History of medical conditions, and history of performing procedures with transmission risk (date, place, type, duration, and frequency),
3. The use of personal protection, i.e., wearing of N95 masks, gloves, and gown, and consistent handwashing.
4. In addition, information will be collected regarding any clinical signs or symptoms in the worker past 3 months, including fever, cough, shortness of breath, or radiographically confirmed pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Age: From 25 to 60 years old
* Department: physicians and nurses from the operating room, critical care department, emergency department, pulmonology department.

Exclusion Criteria:

* pregnant
* Age over 60 years

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be the HCWs at great risk of getting an infection which include those who are in direct contact with respiratory secretions.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Number of IGg seropositive health care workers | single measurement from each person collected over 2 months
  health care workers who have positive IGg in seum

SECONDARY OUTCOMES:
Differentiation between low risk and high risk HCWs | 2 months through out duration of study
  to know positive IGg persons and IGg negative persons to understand risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mukhtar, M.D, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Mizumoto K, Kagaya K, Zarebski A, Chowell G. Estimating the asymptomatic proportion of coronavirus disease 2019 (COVID-19) cases on board the Diamond Princess cruise ship, Yokohama, Japan, 2020. Euro Surveill. 2020 Mar;25(10):2000180. doi: 10.2807/1560-7917.ES.2020.25.10.2000180. PMID 32183930